Brief Title: GER Poses a Potential Risk for Late Complications of BPD

Official Title: Gastroesophageal Reflux Really Pose a Potential Risk for

Late Complications of Bronchopulmonary Dysplasia in Extremely

**Premature Infants** 

Identifiers: NCT03014453

Unique Protocol ID:A333-1

Sponsor: Shengjing Hospital

Investigator: Shucheng Zhang

Official Title: Professor

Affiliation: Shengjing Hospital

Document Date: March 24, 2020

## **Informed Consent Form**

### Research background

Your case will be reported by professor Shucheng ZHANG of Shengjing Hospital of China Medical University.

This study has been approved by the ethical review committee of Shengjing Hospital of China Medical University. This form describes the purpose, process, and method of the study; please take time to review it. If you decide to take part in the study, you will be asked to sign this form.

## Research purposes

Bronchopulmonary dysplasia (BPD) is common in low birth weight infants. Although most of the BPD symptoms improved after a regular treatment in infancy, there are still a few late complications left, such as frequent respiratory symptoms, slower weight gain and even sudden death. These late complications have made so much trouble to the healthcare of BPD infants. How to find the risk factors and to reduce the prevalence of these late symptoms becomes necessary. In this study, a cohort of BPD infants was observed with the late complications obtained by a monthly followed up for 18 months after discharge, the prevalence and risk factors were analyzed via logistic regression, calculating odd ratios (OR) and 95% confidence intervals. As one of the risk factors, GER was verified whether to play a critical role in these late complications.

#### Research process and methods

If you agree to participate in this study, we will number you and establish medical records. In the course of the study, we will need you to agree to take a 24-hour gastric-esophageal pH test, and truthfully report changes in health conditions after discharge from the hospital. Your medical records will be collected, and participants will be followed for 18 months.

#### Research significance

Your case report will help doctors make a diagnosis, and perform treatment. Furthermore, it will provide information for researchers on the late complications of bronchopulmonary dysplasia

# **Privacy policy**

Researchers will protect your privacy.

#### **Statement**

Taking part in this study is completely voluntary. You do not have to participate if you don't want to. You may also leave the study at any time. If you leave the study before it is finished, there will be no penalty, and you will not lose any benefits to which you are otherwise entitled.

## **Signature**

I understand the information printed on this form. My questions so far have been answered. I agree to take part in this study.

Signature

Date